CLINICAL TRIAL: NCT03880058
Title: Safety and Efficacy of SLI-F06 in Wound Healing and Scar Appearance in Pre-Abdominoplasty Surgical Excisions and Post-Operative Scar Appearance In Subjects Undergoing Abdominoplasty
Brief Title: Safety and Efficacy of SLI-F06 in Wound Healing and Scar Appearance
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Scarless Laboratories, Inc. (Industry)
Collaborators: ethica Clinical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SLI-C40-001
Record Dates: First submitted 2019-03-05; First posted 2019-03-19 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Scars
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SLI-F06 (Active Comparator): Drug Product under investigation
  Interventions: Drug: SLI-F06
- Formulation Buffer (Placebo Comparator): Placebo
  Interventions: Drug: Formulation buffer

INTERVENTIONS:
Drug: SLI-F06 — Active treatment
  Other Names: F06-C40
  Arms: SLI-F06
Drug: Formulation buffer — Placebo treatment
  Other Names: Placebo, vehicle
  Arms: Formulation Buffer

SUMMARY:
Multicenter, double-blind study comparing SLI-F06 to vehicle formulation buffer for the improvement in scar appearance and wound strength in routine surgical excisions, as well as post-operative abdominoplasty scar appearance.

DETAILED DESCRIPTION:
The study is divided into 2 parts where Part A is a Phase I safety/proof of concept study of small scars pre-abdominoplasty, and Part B is a Phase IIa study of post-abdominoplasty scars.

In Part A of the study, subjects will have their abdominoplasty site mapped to accommodate a series of excisions depending on pannus size. All excisions to be treated with SLI-F06 will be on one side of the mapped area (i.e., left side or right side) and vehicle treated excisions will be on the other side of the mapped area. At time of abdominoplasty the excision site will be harvested and processed.

In Part B of the study, subjects who complete Part A will be randomly assigned to receive injections of SLI-F06 along one half (left or right) of the abdominoplasty incision and control injections along the other half. The subject will undergo routine wound care and will attend study follow-up visits following abdominoplasty. The entire incision will be treated post-operatively in precisely the same manner.

Duration of study-approximately 26 months.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatient, male or female of any race, 18 years of age or older. Female subjects of childbearing potential must have a negative urine pregnancy test (UPT) at Visit 1a and 1b and practice a reliable method of contraception throughout the study.
2. Seeking or scheduled for standard elective abdominoplasty.
3. Willing to undergo directed excisions and follow-up prior to abdominoplasty and to undergo all follow-up visits after abdominoplasty.
4. Willing to undergo directed excisions under local anesthetic
5. Be able to follow study instructions and likely to complete all required visits.
6. Sign the Institutional Review Board (IRB)-approved Informed Consent Form (ICF), which includes the Photographic Release Form and HIPAA, prior to any study-related procedures being performed.

Exclusion Criteria:

1. Female subjects that are pregnant, breast-feeding, or of childbearing potential and not practicing reliable birth control.
2. Known hypersensitivity or previous allergic reaction to any constituent of the investigational product (IP).
3. History of diabetes mellitus or a Hemoglobin (HgB) A1C greater than 5.7 percent.
4. Morbid obesity (i.e., BMI >40).
5. History of prior abdominal surgery.
6. History of abdominal liposuction, cryolipolysis, focused ultrasound or other fat reduction procedures in or near the anterior abdomen within 12 months of baseline.
7. History of poor or delayed wound healing such as a prior wound dehiscence, chronic wound or leg ulcer.
8. History of or evidence of a genetic collagen disorder such as Ehlers-Danlos syndrome.
9. Operating Physician unable to design an abdominoplasty incision area of at least 25 cm wide by 12 cm tall at the center of the fusiform.
10. The presence of any abnormality of the skin within the area of the proposed abdominoplasty that, in the opinion of the Principal Investigator (PI), could interfere with the excision process or grading of the resultant surgical scar.
11. Use of any restricted concomitant medications/procedures or tobacco/inhaled nicotine products within a restricted time period.
12. Allergy to or intolerance of local anesthetics.
13. Medical or psychiatric conditions that may increase the risk associated with study participation or may interfere with interpretation of study results or compliance of the subject and, in the opinion of the PI, would make the subject inappropriate for study entry.
14. Any personal, familial, employment or financial situation that could impede the subject's ability to attend all study visits and successfully complete the entire clinical study.
15. Clinically significant alcohol or drug abuse, or history of poor cooperation or unreliability.
16. Exposure to any other investigational drug/device within 30 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D. Galiano, MD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Site 1, Chicago, Illinois
  - Site 2, St Louis, Missouri
  - Site 3, Bala-Cynwyd, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Pre and post abdominoplasty scars
Groups:
- All Study Participants: All study participants served as their own control. In Part A, subjects had their abdominoplasty site mapped with equal excisions on left/right of midline to accommodate small (12), medium (14) or large (18) pannus excisions with standardized 3 cm length. In Part B, subjects received injections of SLI-F06 along one half (left/right) of the abdominoplasty incision and control injections along the other half.
  The solution of SLI-F06 or vehicle solution was injected intradermally into BOTH edges of the surgical wound immediately prior to closure (Part A) and before/after closure (Part B). The concentration of SLI-F06 was 25 mg/ml.
  In Part A, a total of 0.4 mL (10 mg) was injected once at each excision site. A total of 0.2 mL (5 mg) was injected along EACH SIDE of the wound edge. As each wound edge was 3 cm in length, 0.05 mL was injected per 0.75 cm of wound edge. The total exposure of SLI-F06 for subjects with small pannus was approximately 60 mg (6 treated excisions), for subjects with a medium pannus approximately 70 mg (7 treated excisions), and for subjects with a large pannus approximately 90 mg (9 treated excisions).
  In Part B of the study, 0.05 mL was injected once per 0.75 cm of wound edge as above. A subject with an incision length of 25 cm (12.5 cm active treatment) was exposed to 41.6 mg of SLI-F06, while subjects with an incision length of 30 cm (15 cm active treatment) or 32 cm (16 cm active treatment) were exposed to 50 mg or 53.3 mg, respectively.
Period: Part A: Pre-abdominoplasty Injections
Arm/Group | All Study Participants
Started | 22; 280 Pre and post abdominoplasty scars
Received SLI-F06 | 22; 140 Pre and post abdominoplasty scars
Received Control | 22; 140 Pre and post abdominoplasty scars
Completed | 22; 280 Pre and post abdominoplasty scars
Not Completed | 0; 0 Pre and post abdominoplasty scars
Period: Part B: Abdominoplasty Injections
Arm/Group | All Study Participants
Started | 21; 21 Pre and post abdominoplasty scars (One patient from Part A did not enroll in Part B)
Received SLI-F06 | 21; 21 Pre and post abdominoplasty scars
Received Control | 21; 21 Pre and post abdominoplasty scars
Completed | 21; 21 Pre and post abdominoplasty scars
Not Completed | 0; 0 Pre and post abdominoplasty scars

BASELINE CHARACTERISTICS:
Population: In Part A, there were 140 treated scars and 140 control scars per subject for a total of 280. In Part B, there was one abdominoplasty incision per patient, with the left or right side receiving treatment or control. Each subject served as their own control.
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Patient and Observer Scar Assessment Scale (POSAS) - PI Assessment
Description: POSAS is an established scale for assessing scar by both the patient and the observer. The overall opinion of the scar is reported on a scale of 1-10, with 1 being normal skin and 10 being the worst scar. Comparisons between treatment groups for efficacy analyses are based on 95% confidence intervals (CI) calculated using mixed models with treatment group as a fixed effect and subject as a random effect to account for multiple observations (i.e., scars) within subject.
Time Frame: Post-excision at Month 3
Population: Part A: Pre-abdominoplasty excisions
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Scars
Arm/Group | SLI-F06 | Formulation Buffer
Number analyzed (Participants) | 22 | 22
Number analyzed (Scars) | 140 | 140
score on a scale | 4.4 (1.7) | 4.5 (1.7)

2. Primary Outcome: Patient and Observer Scar Assessment Scale (POSAS) - PI Assessment
Description: as for outcome 1
Time Frame: Post-abdominoplasty at Month 12
Population: Part B: Abdominoplasty incisions
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Scars
Arm/Group | SLI-F06 | Formulation Buffer
Number analyzed (Participants) | 21 | 21
Number analyzed (Scars) | 21 | 21
score on a scale | 1.6 (1.7) | 1.7 (1.7)

ADVERSE EVENTS:
Time Frame: Subjects were assessed at Visit 4a (Day 29), Visit 5a (Day 57 - Group 2 only), Visit 6a (Day 85 - Group 1 only), Visits 3b-12b (M1-3, 6, 9, 12, 15, 18, 21 and 24 at study exit).
Description: No difference in definition
  Systematic Assessment: Subjects were questioned for the occurrence of any new or worsening signs or symptoms at each visit. Safety laboratory tests were conducted at select study visits. Clinically significant adverse events were reported.
Arm/Group | SLI-F06 | Formulation Buffer
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 3/22 | 3/22
Other Adverse Events (participants affected / at risk) | 14/22 | 14/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SLI-F06 (N=22) | Formulation Buffer (N=22)
Pulmonary embolism (Vascular disorders) | 1 (1) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SLI-F06 (N=22) | Formulation Buffer (N=22)
Seroma drainage (Surgical and medical procedures) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dermoid cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Synovial cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Allergy to surgical sutures (General disorders) | 1 (1) | 1 (1)
Tension headache (Nervous system disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Drain site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Incision site hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dermatitis allergic (Immune system disorders) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT03880058/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT03880058/SAP_001.pdf